CLINICAL TRIAL: NCT00032643
Title: CSP #526 - A Thyroid Hormone Analog to Fight Heart Failure: Phase II Trial (DITPA)
Brief Title: A Thyroid Hormone Analog to Fight Heart Failure: Phase II Trial (DITPA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding support withdrawn (much slower than expected enrollment)
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Masking: Double
Other Study IDs: 526
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: DITPA

INTERVENTIONS:
Drug: DITPA

SUMMARY:
Congestive heart failure (CHF) affects 4-5 million Americans, and its prevalence is predicted to increase over the next few decades. Thyroid hormone has unique actions which make it a novel and potentially useful agent for treatment of CHF. Due to possible adverse affects of thyroid hormone, there is interest in developing analogs with fewer undesirable side effects. 3,5- diiodothyropropionic acid (DITPA) has been shown to improve diastolic function in both animal models and a recently completed double-blind placebo controlled trial in 19 humans.

The goal of the proposed Phase II study is to show safety and demonstrate a medication of efficacy of DITPA needed in patients with CHF. This study is a prerequisite for a larger Phase III trial which would determine whether mortality is improved with DITPA. To better define the appropriate doses, prior to the Phase II study we will conduct an initial pharmacokinetic study.

DETAILED DESCRIPTION:
Intervention: After enrollment, patients receive a clinical assessment, echocardiogram and laboratory studies. Then, each patient receives treatment with one of two doses of 3,5-diiodothyropropionic acid (DITPA) or placebo for six months.

Primary hypothesis: DITPA will improve cardiovascular function and clinical status in patients with moderately severe heart failure and be similar to placebo on safety measures.

Secondary hypothesis:

Primary Outcomes: 1. Composite endpoint composed of cardiovascular mortality/morbidity, change in NYHA class and change in global assessment, and 2. safety.

Study Abstract: Congestive heart failure (CHF) affects 4-5 million Americans, and its prevalence is predicted to increase over the next few decades. Thyroid hormone has unique actions which make it a novel and potentially useful agent for treatment of CHF. Due to possible adverse effects of thyroid hormone, there is interest in developing analogs with fewer undesirable side effects. DITPA has been shown to improve diastolic function in both animal models and a recently completed double-blind placebo controlled trial in 19 humans.

The goal of the proposed Phase II study is to define the dose of DITPA needed to achieve hemodynamic improvement in patients with CHF. This study is a prerequisite for a larger Phase III trial which would determine whether mortality is improved with DITPA. To better define the appropriate doses, prior to the Phase II study we will conduct an initial pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION

To be enrolled, patients must:

1. be veterans,
2. have moderately severe CHF (NYHA class II, III or IV),
3. be 18 or older,
4. not have clinically important renal, hepatic or hematological disorders or clinically significant abnormal laboratory findings,
5. not have a pre-existing thyroid disease,
6. not have anemia (hematocrit less than 30%),
7. not have chronic pulmonary disease that limits exercise tolerance or requires use of chronic bronchodilator therapy or steroids,
8. be able to walk on the level for 6 minutes,
9. not have hemodynamically significant pericardial disease,
10. not have angina pectoris severe enough to require frequent administration of sublingual nitroglycerin,
11. not have acute myocardial infarction within 6 months of screening,
12. not have inoperable aortic stenosis,
13. not have symptomatic ventricular arrhythmias or ventricular arrhythmia requiring pharmacological therapy,
14. not have implanted cardioverter defibrillator,
15. not be taking amiodarone,
16. not have demonstrated non-compliance with prior medical regimes;
17. not be on an investigational drug,
18. not have a medical condition that, in the investigator's opinion, would make the patient ineligible,
19. not have an allergy to iodine or shellfish,
20. not be in sinus rhythm,
21. not be of childbearing potential,
22. have an ejection fraction greater than 40%.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Goldman, MD, Study Chair — Southern Arizona VA Health Care System
Locations (7):
- United States (7):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas